CLINICAL TRIAL: NCT07143747
Title: PAXT: Pulmonary Imaging of Mild Asthma Using 129Xe MRI and Tc-99-Labeled-Carbon-Imaging (Tc99CImaging)
Acronym: PAXT
Status: Not yet recruiting | Type: Observational
Sponsor: Dr. Grace Parraga (Other)
Collaborators: Cyclomedica Australia PTY Limited (Industry)
Responsible Party: Sponsor-Investigator, Dr. Grace Parraga, Professor, Western University, Canada
Organization: Western University, Canada (Other)
Other Study IDs: ROB0055
Record Dates: First submitted 2025-08-08; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Mild Asthma
Keywords: Hyperpolarized 129Xe MRI; Technegas Ventilation Imaging; Pulmonary Function Testing; Mild Asthma; Ventilation Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mild Asthma
  Interventions: Other: Hyperpolarized 129Xe MRI; Other: Tc-99m Technegas Ventilation Imaging

INTERVENTIONS:
Other: Hyperpolarized 129Xe MRI — Inhalation of hyperpolarized 129Xe gas followed by breath-hold MRI for ventilation imaging.
Other: Tc-99m Technegas Ventilation Imaging — Inhalation of Tc-99m-labeled carbon aerosol (Technegas) followed by SPECT imaging to assess lung ventilation.

SUMMARY:
The goal of this observational study is to better understand how asthma affects the lungs in young adults (ages 17-35) with mild asthma. The main questions it aims to answer are:

* Can advanced imaging detect abnormal airway function in people with mild asthma?
* Do changes in ventilation imaging correlate with asthma symptoms or quality of life? Researchers will compare hyperpolarized xenon-129 MRI and Technegas (Tc-99m) imaging to see if these techniques reveal more detailed lung abnormalities than standard lung function tests.

Participants will:

* Complete a single 2-hour visit
* Undergo two types of lung imaging: Hyperpolarized xenon-129 MRI (to visualize how air moves in the lungs), Technegas (Tc-99m) imaging (to assess airflow using nuclear medicine)
* Perform spirometry and other breathing tests
* Answer questionnaires about asthma symptoms and quality of life This study is designed to improve our understanding of subtle changes in lung function that may not be detected by standard tests in people with mild asthma. The findings may lead to better diagnostic tools and more personalized treatment strategies in the future.

DETAILED DESCRIPTION:
This is a single centre, study in university-aged participants diagnosed with mild asthma as indicated by a prescription for a short acting bronchodilator for use as needed.

Each participant will participate in one research study visit which includes pre- and post- bronchodilator (BD) spirometry, plethysmography, oscillometry, 129Xe MRI as well as pre-BD ultra-low dose chest CT, Tc99CImaging, blood CBC, sputum induction, as well as completion of the ACQ and AQLQ questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study must meet all of the following criteria:

1. Participant diagnosed with mild (GINA1) asthma by physician
2. Participant understands study procedures and is willing to participate in the study as indicated by the participant's signature
3. Provision of written, informed consent prior to any study specific procedures
4. Males and females 17 to 35 years of age
5. Women of childbearing potential (after menarche) must ensure that they are using an effective form of birth control for at least 2 months prior to each imaging visit. Examples of effective birth control include:

   1. True sexual abstinence
   2. A vasectomized sexual partner
   3. Implanon®
   4. Female sterilization by tubal occlusion
   5. Effective intrauterine device (IUD)/levonogestrel intrauterine system (IUS)
   6. Depo-Provera™ injections
   7. Oral contraceptive
   8. Evra Patch™
   9. Nuvaring™

Exclusion Criteria:

Participants fulfilling any of the following criteria are not eligible for inclusion in this study:

1. Participant has an implanted mechanically, electrically, or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) (at the discretion of the MRI Technologist)
2. In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, CT, or Tc99CImaging, such as severe claustrophobia
3. Participants who are pregnant, breastfeeding or have a positive pregnancy test at initial screening visit
4. Participant is unable to perform spirometry or plethysmography maneuvers
5. Participant is unable to perform MRI and CT breath-hold maneuvers

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be young adults aged 17 to 35 years with physician-diagnosed mild asthma, consistent with Global Initiative for Asthma (GINA) Step 1 criteria. All participants will be prescribed short-acting bronchodilators for as-needed use only and will have no regular controller medication use. Eligible individuals must be otherwise healthy, non-smokers (or with ≤5 pack-year history and no smoking in the past year), and free from other chronic respiratory diseases. Participants will be recruited from the general population and will undergo a single, comprehensive imaging and lung function assessment visit.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Measure 129Xe and Tc99C Imaging ventilation defects qualitatively and quantitatively in participants diagnosed and treated as "mild" asthma. | 1 baseline visit for pre- and post-bronchodilator imaging assessments
  Ventilation defects will be assessed using 129Xe MRI and Tc-99m Technegas SPECT imaging. Measurements will include ventilation defect percentage (VDP) and visual scoring to evaluate ventilation abnormalities in participants with mild asthma.

SECONDARY OUTCOMES:
Evaluate the relationships of MRI and Tc99CImaging ventilation defects with ACQ, oscillometry (R5-19) and FEV1 | 1 baseline visit
  In this exploratory study, we hypothesize that there will be significant relationships between ventilation abnormalities and oscillometry as well as FEV1 and asthma control questionnaire (ACQ) score.

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No